CLINICAL TRIAL: NCT00519662
Title: Phase 1 Open-Label Multicenter, Dose-Escalating, Clinical Study of the Safety, Tolerability, and Pharmacokinetic and Pharmacodynamic Profiles of SNS-314, a Novel Aurora Kinase Inhibitor, Administered to Patients With Advanced Solid Tumors
Brief Title: Safety and Tolerability Study of SNS-314 for Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sunesis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPO-0011
Record Dates: First submitted 2007-08-20; First posted 2007-08-22 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Advanced Solid Tumors
Keywords: Solid; Tumors; Advanced
MeSH Terms: conditions — Neoplasms | interventions — SNS 314

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dose escalating cohorts of SNS-314 (Experimental): Sequential groups, starting at a dose of 30 mg/m2, will be escalated according to identification of dose limiting toxicities against various criteria. Doses escalated by doubling the dose until the first observation of clinically significant Grade 2 or greater toxicity related to SNS-314 injection. Results in dosing increments of 67%, 50%, 40%, 33%, and subsequently 25% based on modified Fibonacci schema.
  Interventions: Drug: SNS-314

INTERVENTIONS:
Drug: SNS-314 — Stage 1 - Escalating doses of SNS-314 Injection on days 1, 8 and 15
  Stage 2 - Same as stage 1 except SNS-314 Injection is administered at the maximum tolerated dose established in stage 1

SUMMARY:
This is a study to assess the safety and tolerability of SNS-314 in advanced solid tumors in humans.

DETAILED DESCRIPTION:
Other objectives of this study include measuring pharmacokinetics (how long the drug can be measured in the blood).

ELIGIBILITY:
Inclusion Criteria:

* Advanced solid tumor and that is measurable by a scan

Exclusion Criteria:

* Uncontrolled or untreated central nervous system metastases
* Cerebrovascular accident/transient ischemic attack up to 6 months before Cycle 1 Day 1
* Any of the following cardiac conditions:
* History of myocardial infarction, acute coronary syndromes up to 12 weeks before Cycle 1 Day 1
* Class III or IV heart failure up to 6 months before Cycle 1 Day 1
* Baseline heart rate corrected QT interval (QTc)> 450 msec
* History of ventricular arrhythmias up to 6 months before Cycle 1 Day 1
* Use of medications that prolong the QTc interval and are associated with Torsades de Pointe (TdP)
* Previous cancer treatment up to 21 days before first dose
* Any investigational therapy up to 28 days before Cycle 1 Day 1
* Known allergy to cyclodextrins

Please note: There are additional inclusion/exclusion criteria for this study. Please contact the study center for additional information and to determine if all study criteria are met.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2007-08; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
To assess the safety and tolerability of SNS-314 | 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Michelson, MD, Study Director — Sunesis Pharmaceuticals
Locations (4):
- United States (4):
  - University of Alabama, Birmingham, Birmingham, Alabama
  - Stanford University Medical Center, Stanford, California
  - University of New Mexico, Albuquerque, New Mexico
  - Duke University, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No